CLINICAL TRIAL: NCT04762537
Title: Surmounting Withdrawal to Initiate Fast Treatment With Naltrexone: Improving the Real-World Effectiveness of Injection Naltrexone for Opioid Use Disorder (SWIFT)
Brief Title: Surmounting Withdrawal to Initiate Fast Treatment With Naltrexone
Acronym: SWIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Principal Investigator, Adam Bisaga, Professor of Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTN-0097; UG1DA013035-19 (NIH)
Record Dates: First submitted 2021-01-21; First posted 2021-02-21 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: The proposed study is an open-label, multi-center, stepped-wedge cluster randomized trial. As part of the stepped-wedge design proposed for this trial, one site, randomly chosen, will start implementing the Rapid procedure (RP) and will remain in this arm for the rest of the study. The next 4 sites randomly chosen will first implement the Standard procedure (SP), to establish the within-site comparison condition, and then at selected staggered time-points (steps) will switch to implementing only the RP. The 6th site (after 5 sites have been randomized to RP) will remain in the SP procedure arm throughout the whole duration of the study. Implementation of RP at study sites will be staggered by 14 weeks and the order in which sites will cross-over from SP to RP will be randomly chosen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Induction Method (Active Comparator): The Standard Method (13-day long) includes 5-days of buprenorphine taper followed by 7-day washout period
  Interventions: Other: Standard Induction Procedure (SP)
- Rapid Induction Method (Experimental): The Rapid Method includes one day of buprenorphine followed by a day of washout and 3-4 days of oral naltrexone titration with adjunctive medications
  Interventions: Other: Rapid Induction Procedure (RP)

INTERVENTIONS:
Other: Standard Induction Procedure (SP) — SP includes stabilization on buprenorphine (6-8 mg) on Day 1 followed by a taper over the subsequent 4 days. After the completion of buprenorphine taper, participants will enter a washout period of at least 8 days. On the last day of the washout period, participants will be evaluated for eligibility to receive XR-NTX injection. Once found eligible, an XR-NTX injection will be given.
  Arms: Standard Induction Method
Other: Rapid Induction Procedure (RP) — RP includes 1 day of buprenorphine 6-8 mg, followed by a day of washout and 4 days of oral naltrexone titration. If the participant is able to tolerate the last dose of the naltrexone titration, an XR-NTX injection will be given
  Arms: Rapid Induction Method

SUMMARY:
This study compares two methods of initiating treatment with extended-release naltrexone (XR-NTX) when implemented at community-based inpatient or residential programs. The primary goal of this hybrid effectiveness-implementation study is to determine whether the Rapid Method (5-7 day long) is non-inferior to a Standard Method (13-day long) on the primary effectiveness outcome of successful initiation of XR-NTX (receiving the first injection). Secondary objectives include comparing Rapid versus Standard method on: time from admission to first dose of XR-NTX and time to dropout, craving, withdrawal severity, retention, abstinence, and safety measures, as measured during the inpatient induction process and the first two months of post-induction XR-NTX maintenance. Other exploratory outcomes include predictors of initiation success, and economic analyses. The implementation goal is to operationalize an implementation facilitation strategy that will be used to train clinical sites on the XR-NTX initiation method, to capture fidelity to the rapid induction process, and to study barriers and facilitators to implementation and refine the implementation facilitation strategy accordingly.

DETAILED DESCRIPTION:
The overarching objective of the SWIFT trial (CTN-0097) is to foster widespread adoption of a regimen for rapid initiation of treatment with extended-release injection naltrexone (XR-NTX) at inpatient or residential Community Treatment Programs (CTPs). If widely adopted, such a regimen would have a substantial public health impact by expanding medication treatment options offered to patients with OUD to include XR-NTX.

In multi-site, randomized (subject level) trials, XR-NTX, once initiated, has been found to have similar effectiveness to sublingual buprenorphine on clinical outcomes of retention in treatment and abstinence from opioids. However, initiation of naltrexone often involves a significant (up to 2 weeks) delay, which is a clinical hurdle that impedes the widespread adoption of XR-NTX as a treatment option. Initiation of naltrexone in patients actively using opioids requires that a patient be detoxified first, and the official prescribing information for XR-NTX recommends an additional 7- to 10-day waiting period after last dose of opioid before administering XR-NTX. This standard initiation regimen, involving a brief period of agonist, usually buprenorphine, taper followed by a 7- to 10-day waiting period, takes approximately two weeks. During this time, patients are vulnerable to drop out and relapse; further, this waiting period is problematic in the face of funding restrictions on the duration of inpatient stays. In a single-site randomized trial, a Rapid naltrexone induction method utilizing minimal buprenorphine, non-opioid medications to treat withdrawal symptoms, and upward titration of oral naltrexone starting with small doses, XR-NTX initiation was accomplished in 5 to 7 days and was found superior to the standard 14-day approach on the proportion of patients initiating XR-NTX.

The primary goal of this hybrid effectiveness-implementation study is to determine whether the Rapid method of initiating treatment with XR-NTX is non-inferior to a standard method on the primary effectiveness outcome of successful initiation of XR-NTX (receiving the first injection) when implemented at community-based inpatient or residential programs. Secondary objectives include comparing rapid versus standard method of XR-NTX initiation on: time from admission to first dose of XR-NTX and time to dropout, craving, withdrawal severity, retention, abstinence, and safety measures, as measured during the inpatient initiation process and the first two months post XR-NTX induction. Other exploratory outcomes include predictors of initiation success, and economic analyses. The implementation goal is to operationalize an implementation facilitation strategy that will be used to train clinical sites on the XR-NTX initiation method, to capture fidelity to the rapid induction process, and to study barriers and facilitators to implementation and refine the implementation facilitation strategy accordingly.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Meets current Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for opioid use disorder.
3. Seeking treatment for opioid use disorder, willing to accept treatment with XR- NTX and, in the judgment of the treating physician, is a good candidate for naltrexone- based treatment.
4. Willing and able to provide written informed consent.
5. Able to speak English sufficiently to understand the study procedures and provide written informed consent to participate in the study.
6. If female of childbearing potential, willing to practice an effective method of birth control for the duration of participation in the study.

Exclusion Criteria:

1. Serious medical, psychiatric or substance use disorder that, in the opinion of the study physician, would make a detoxification and naltrexone initiation, or maintenance treatment with XR-NTX, hazardous (relative contra-indications) or requires a different level of care. Examples include:

1. Disabling or terminal medical illness (e.g., uncompensated heart failure, severe acute hepatitis, cirrhosis or end-stage liver disease) as assessed by medical history and/or review of systems.
2. Severe, untreated or inadequately treated mental disorder (e.g., active psychosis, uncontrolled manic-depressive illness) as assessed by history and/or clinical interview.
3. Current severe alcohol, benzodiazepine, or other depressant or sedative hypnotic use likely to require a complicated medical detoxification (routine alcohol and sedative detoxifications may be included).
4. Suicidal or homicidal ideation that requires immediate attention. Known allergy or sensitivity to buprenorphine, naloxone, naltrexone, polylactide-co-glycolide, carboxymethylcellulose, or other components of the Vivitrol® diluent.

   3. Maintenance treatment with methadone. 4. Maintenance treatment with buprenorphine unless the patient is determined to have a poor treatment response (in the form of buprenorphine non-adherence with or without the use of illicit opioids), warranting change to XR-NTX treatment.

   5. Presence of pain of sufficient severity as to require ongoing pain management with opioids.

   6. Circumstances (legal, personal, occupational) that would threaten the feasibility of XR- NTX treatment or make another treatment (e.g. buprenorphine or methadone) a better choice.

   7. Are currently in jail, prison or other overnight facility as required by court of law or have pending legal action that could prevent participation in study activities.

   8. If female, currently pregnant or breastfeeding, or planning on conception. 9. Body habitus that, in the judgment of the study physician, precludes safe intramuscular injection of XR-NTX (e.g., BMI>40, excess fat tissue over the buttocks, emaciation).

   10. Admitted to the inpatient detoxification or residential rehabilitation unit more than 3 days prior to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Aspire Health Partners, Orlando, Florida
  - Avery Road Treatment Center, Rockville, Maryland
  - Gibson Recovery Center, Inc., Cape Girardeau, Missouri
  - Stony Brook Eastern Long Island Hospital, Greenport, New York
  - Adapt, Roseburg, Oregon
  - Nexus Recovery Center, Inc., Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the National Institutes of Health (NIH) Data Sharing Policy and Implementation Guidance (https://grants.nih.gov/grants/policy/data_sharing/data_sharing_guidance.htm) and (for HEAL-funded studies) the Helping to End Addiction Long-term (HEAL) Public Access and Data Sharing Policy (https://www.nih.gov/research-training/medical-research-initiatives/heal-initiative/research/heal-public-access-data-sharing-policy).
  Primary data for this study will be available to the public in the National Institute on Drug Abuse (NIDA) data repository. For more details on data sharing please visit https://datashare.nida.nih.gov/.
  The primary outcome(s) publication will be included along with study underlying primary data in the data share repository, and it will also be deposited in PubMed Central http://www.pubmedcentral.nih.gov/ per NIH Policy (http://publicaccess.nih.gov/).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
URL: https://datashare.nida.nih.gov

REFERENCES:
- [Result] Sullivan M, Bisaga A, Pavlicova M, Choi CJ, Mishlen K, Carpenter KM, Levin FR, Dakwar E, Mariani JJ, Nunes EV. Long-Acting Injectable Naltrexone Induction: A Randomized Trial of Outpatient Opioid Detoxification With Naltrexone Versus Buprenorphine. Am J Psychiatry. 2017 May 1;174(5):459-467. doi: 10.1176/appi.ajp.2016.16050548. Epub 2017 Jan 10. PMID 28068780
- [Derived] Shulman M, Greiner MG, Tafessu HM, Opara O, Ohrtman K, Potter K, Hefner K, Jelstrom E, Rosenthal RN, Wenzel K, Fishman M, Rotrosen J, Ghitza UE, Nunes EV, Bisaga A. Rapid Initiation of Injection Naltrexone for Opioid Use Disorder: A Stepped-Wedge Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e249744. doi: 10.1001/jamanetworkopen.2024.9744. PMID 38717773
- [Derived] Greiner MG, Shulman M, Opara O, Potter K, Voronca DC, Tafessu HM, Hefner K, Hamilton A, Scheele C, Ho R, Dresser L, Jelstrom E, Fishman M, Ghitza UE, Rotrosen J, Nunes EV, Bisaga A. Surmounting Withdrawal to Initiate Fast Treatment with Naltrexone (SWIFT): A stepped wedge hybrid type 1 effectiveness-implementation study. Contemp Clin Trials. 2023 May;128:107148. doi: 10.1016/j.cct.2023.107148. Epub 2023 Mar 15. PMID 36931426

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 451 participants were found eligible at pre-screening, 32 of which did not meet eligibility criteria at screening. Of the 419 participants determined eligible at screening, 4 withdrew interest in participation or left prior to completion of screening and initiation of enrollment. The total remaining 415 were enrolled in one of the study treatment arms.
Units Other Than Participants: Sites
Groups:
- Site 1: Rapid Procedure for Duration of Study (70 Weeks): The Rapid Method includes one day of buprenorphine followed by a day of washout and 3-4 days of oral naltrexone titration with adjunctive medications
  Rapid Induction Procedure (RP): RP includes 1 day of buprenorphine 6-8 mg, followed by a day of washout and 4 days of oral naltrexone titration. If the participant is able to tolerate the last dose of the naltrexone titration, an XR-NTX injection will be given
- Site 2: 14 Weeks of Standard Procedure, Followed by 56 Weeks of Rapid Procedure: The Standard Method (13-day long) includes 5-days of buprenorphine taper followed by 7-day washout period
  Standard Induction Procedure (SP): SP includes stabilization on buprenorphine (6-8 mg) on Day 1 followed by a taper over the subsequent 4 days. After the completion of buprenorphine taper, participants will enter a washout period of at least 8 days. On the last day of the washout period, participants will be evaluated for eligibility to receive XR-NTX injection. Once found eligible, an XR-NTX injection will be given.
  --
  The Rapid Method includes one day of buprenorphine followed by a day of washout and 3-4 days of oral naltrexone titration with adjunctive medications
  Rapid Induction Procedure (RP): RP includes 1 day of buprenorphine 6-8 mg, followed by a day of washout and 4 days of oral naltrexone titration. If the participant is able to tolerate the last dose of the naltrexone titration, an XR-NTX injection will be given
- Site 3: 28 Weeks of Standard Procedure, Followed by 42 Weeks of Rapid Procedure; Site 4: 42 Weeks of Standard Procedure, Followed by 28 Weeks of Rapid Procedure; Site 5: "Standard Procedure for 56 Weeks, Followed by 14 Weeks of Rapid Procedure: The Standard Method (13-day long) includes 5-days of buprenorphine taper followed by 7-day washout period
  Standard Induction Procedure (SP): SP includes stabilization on buprenorphine (6-8 mg) on Day 1 followed by a taper over the subsequent 4 days. After the completion of buprenorphine taper, participants will enter a washout period of at least 8 days. On the last day of the washout period, participants will be evaluated for eligibility to receive XR-NTX injection. Once found eligible, an XR-NTX injection will be given.
  The Rapid Method includes one day of buprenorphine followed by a day of washout and 3-4 days of oral naltrexone titration with adjunctive medications
  Rapid Induction Procedure (RP): RP includes 1 day of buprenorphine 6-8 mg, followed by a day of washout and 4 days of oral naltrexone titration. If the participant is able to tolerate the last dose of the naltrexone titration, an XR-NTX injection will be given
- Site 6: Standard Procedure for Duration of the Study (70 Weeks): The Standard Method (13-day long) includes 5-days of buprenorphine taper followed by 7-day washout period
  Standard Induction Procedure (SP): SP includes stabilization on buprenorphine (6-8 mg) on Day 1 followed by a taper over the subsequent 4 days. After the completion of buprenorphine taper, participants will enter a washout period of at least 8 days. On the last day of the washout period, participants will be evaluated for eligibility to receive XR-NTX injection. Once found eligible, an XR-NTX injection will be given.
Period: Step 1 (Weeks 0-14)
Arm/Group | Site 1: Rapid Procedure for Duration of Study (70 Weeks) | Site 2: 14 Weeks of Standard Procedure, Followed by 56 Weeks of Rapid Procedure | Site 3: 28 Weeks of Standard Procedure, Followed by 42 Weeks of Rapid Procedure | Site 4: 42 Weeks of Standard Procedure, Followed by 28 Weeks of Rapid Procedure | Site 5: "Standard Procedure for 56 Weeks, Followed by 14 Weeks of Rapid Procedure | Site 6: Standard Procedure for Duration of the Study (70 Weeks)
Started | 14; 1 Sites | 14; 1 Sites | 6; 1 Sites | 25; 1 Sites | 15; 1 Sites | 8; 1 Sites
Completed | 7; 1 Sites | 6; 1 Sites | 1; 1 Sites | 6; 1 Sites | 12; 1 Sites | 1; 1 Sites
Not Completed | 7; 0 Sites | 8; 0 Sites | 5; 0 Sites | 19; 0 Sites | 3; 0 Sites | 7; 0 Sites
Period: Step 2 (Weeks 14-28)
Arm/Group | Site 1: Rapid Procedure for Duration of Study (70 Weeks) | Site 2: 14 Weeks of Standard Procedure, Followed by 56 Weeks of Rapid Procedure | Site 3: 28 Weeks of Standard Procedure, Followed by 42 Weeks of Rapid Procedure | Site 4: 42 Weeks of Standard Procedure, Followed by 28 Weeks of Rapid Procedure | Site 5: "Standard Procedure for 56 Weeks, Followed by 14 Weeks of Rapid Procedure | Site 6: Standard Procedure for Duration of the Study (70 Weeks)
Started | 7; 1 Sites | 25; 1 Sites | 9; 1 Sites | 24; 1 Sites | 13; 1 Sites | 6; 1 Sites
Completed | 4; 1 Sites | 19; 1 Sites | 5; 1 Sites | 7; 1 Sites | 7; 1 Sites | 3; 1 Sites
Not Completed | 3; 0 Sites | 6; 0 Sites | 4; 0 Sites | 17; 0 Sites | 6; 0 Sites | 3; 0 Sites
Period: Step 3 (Weeks 28-42)
Arm/Group | Site 1: Rapid Procedure for Duration of Study (70 Weeks) | Site 2: 14 Weeks of Standard Procedure, Followed by 56 Weeks of Rapid Procedure | Site 3: 28 Weeks of Standard Procedure, Followed by 42 Weeks of Rapid Procedure | Site 4: 42 Weeks of Standard Procedure, Followed by 28 Weeks of Rapid Procedure | Site 5: "Standard Procedure for 56 Weeks, Followed by 14 Weeks of Rapid Procedure | Site 6: Standard Procedure for Duration of the Study (70 Weeks)
Started | 10; 1 Sites | 23; 1 Sites | 12; 1 Sites | 15; 1 Sites | 13; 1 Sites | 7; 1 Sites
Completed | 2; 1 Sites | 14; 1 Sites | 9; 1 Sites | 5; 1 Sites | 4; 1 Sites | 3; 1 Sites
Not Completed | 8; 0 Sites | 9; 0 Sites | 3; 0 Sites | 10; 0 Sites | 9; 0 Sites | 4; 0 Sites
Period: Step 4 (Weeks 42-56)
Arm/Group | Site 1: Rapid Procedure for Duration of Study (70 Weeks) | Site 2: 14 Weeks of Standard Procedure, Followed by 56 Weeks of Rapid Procedure | Site 3: 28 Weeks of Standard Procedure, Followed by 42 Weeks of Rapid Procedure | Site 4: 42 Weeks of Standard Procedure, Followed by 28 Weeks of Rapid Procedure | Site 5: "Standard Procedure for 56 Weeks, Followed by 14 Weeks of Rapid Procedure | Site 6: Standard Procedure for Duration of the Study (70 Weeks)
Started | 15; 1 Sites | 32; 1 Sites | 4; 1 Sites | 23; 1 Sites | 18; 1 Sites | 12; 1 Sites
Completed | 11; 1 Sites | 19; 1 Sites | 2; 1 Sites | 14; 1 Sites | 8; 1 Sites | 1; 1 Sites
Not Completed | 4; 0 Sites | 13; 0 Sites | 2; 0 Sites | 9; 0 Sites | 10; 0 Sites | 11; 0 Sites
Period: Step 5 (Weeks 56-70)
Arm/Group | Site 1: Rapid Procedure for Duration of Study (70 Weeks) | Site 2: 14 Weeks of Standard Procedure, Followed by 56 Weeks of Rapid Procedure | Site 3: 28 Weeks of Standard Procedure, Followed by 42 Weeks of Rapid Procedure | Site 4: 42 Weeks of Standard Procedure, Followed by 28 Weeks of Rapid Procedure | Site 5: "Standard Procedure for 56 Weeks, Followed by 14 Weeks of Rapid Procedure | Site 6: Standard Procedure for Duration of the Study (70 Weeks)
Started | 6; 1 Sites | 13; 1 Sites | 5; 1 Sites | 12; 1 Sites | 24; 1 Sites | 5; 1 Sites
Completed | 4; 1 Sites | 10; 1 Sites | 3; 1 Sites | 11; 1 Sites | 12; 1 Sites | 1; 1 Sites
Not Completed | 2; 0 Sites | 3; 0 Sites | 2; 0 Sites | 1; 0 Sites | 12; 0 Sites | 4; 0 Sites

BASELINE CHARACTERISTICS:
Population: Baseline population includes participants who were enrolled in the study in either the Standard or Rapid treatment arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Induction Method | Rapid Induction Method | Total
Number analyzed (Participants) | 190 | 225 | 415
Age, Categorical [Count of Participants; unit: Participants] — Participants younger than 18 were ineligible to participate in the study.
  Participants
    <=18 years | 0 | 2 | 2
    Between 18 and 65 years | 22 | 24 | 46
    >=65 years | 168 | 199 | 367
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 133 | 210
  Male | 113 | 92 | 205
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Both race and ethnicity were collected independently in this study via participant self-report in pre-determined categories. Ethnicity will be reported here.
  Ethnicity categories include: Hispanic or Latino, Not Hispanic or Latino, Don't know
  Participants
    Hispanic or Latino | 38 | 53 | 91
    Not Hispanic or Latino | 147 | 172 | 319
    Unknown or Not Reported | 5 | 0 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Both race and ethnicity were collected independently in this study via participant self-report in pre-determined categories. Race will be reported here.
  Race categories include: American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Pacific Islander, White, Other, Multiracial, Don't know, Refused to answer
  Participants
    American Indian or Alaska Native | 4 | 1 | 5
    Asian | 4 | 2 | 6
    Black or African American | 28 | 26 | 54
    Native Hawaiian or Pacific Islander | 1 | 1 | 2
    White | 115 | 175 | 290
    Other | 12 | 11 | 23
    Multiracial | 16 | 6 | 22
    Don't Know | 10 | 2 | 12
    Refused to Answer | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 190 | 225 | 415
Education Completed [Count of Participants; unit: Participants] — Categories of completed education milestones collected via participant self-report.
  Participants
    Less than high school diploma | 39 | 49 | 88
    High school graduate | 58 | 69 | 127
    GED or equivalent | 24 | 34 | 58
    Some college, no degree | 38 | 40 | 78
    Associate's degree: occupational, technical, or vocational program | 11 | 9 | 20
    Associate's degree: academic program | 11 | 8 | 19
    Bachelor's degree | 4 | 7 | 11
    Master's degree | 3 | 3 | 6
    Professional school degree | 0 | 0 | 0
    Doctoral degree | 0 | 0 | 0
    Don't know | 2 | 6 | 8
Marital Status [Count of Participants; unit: Participants] — Marital status collected via participant self-report
  Participants
    Married | 15 | 16 | 31
    Widowed | 4 | 7 | 11
    Divorced | 23 | 28 | 51
    Separated | 15 | 15 | 30
    Never married | 112 | 121 | 233
    Living with partner | 16 | 28 | 44
    Don't know | 4 | 10 | 14
    Refused | 1 | 0 | 1
Sexual-Orientation [Count of Participants; unit: Participants] — Sexual orientation collected via participant self-report
  Participants
    Missing | 23 | 21 | 44
    Heterosexual or straight | 146 | 173 | 319
    Gay or lesbian | 2 | 4 | 6
    Bisexual | 15 | 24 | 39
    Queer | 2 | 0 | 2
    Not sure | 1 | 2 | 3
    Something else | 1 | 1 | 2
Employment [Count of Participants; unit: Participants] — Collected via participant self-report
  Participants
    Working now | 50 | 52 | 102
    Only temporarily laid off, sick leave, or maternity leave | 5 | 15 | 20
    Looking for work, unemployed | 121 | 140 | 261
    Retired | 1 | 0 | 1
    Disabled permanently or temporarily | 6 | 4 | 10
    Keeping house | 3 | 12 | 15
    Student | 1 | 1 | 2
    Other | 3 | 1 | 4
Location participant spent the night before coming to the unit [Count of Participants; unit: Participants] — Collected via participant self-report
  Participants
    Missing | 22 | 32 | 54
    Own apartment, room or house - subsidized, for example Section 8 or living in public housing | 9 | 3 | 12
    Own apartment, room or house - not subsidized | 47 | 84 | 131
    Someone else's apartment, room or house | 66 | 65 | 131
    Hotel, SRO, or boarding home | 17 | 8 | 25
    Halfway house, residential treatment program (focus: establishing sobriety) | 1 | 3 | 4
    Transitional housing (focus: movement into permanent housing) | 1 | 2 | 3
    Institution (hospital, nursing home, etc.) | 4 | 3 | 7
    Homeless shelter | 4 | 1 | 5
    Outdoors/street, abandoned/public building, vehicle, or other place not meant for human habitation | 11 | 11 | 22
    Detox | 1 | 1 | 2
    Other - homeless | 3 | 3 | 6
    Other - stable housing | 1 | 4 | 5
    Other | 3 | 5 | 8
First COWS Score on Day 1 of admission [Mean (Standard Deviation); unit: units on a scale] — COWS (Clinical Opioid Withdrawal Scale) measures withdrawal symptom severity with a 0-48 point scale, with 0 points indicating no symptoms are observed, and 48 points indicating maximum severity.
  There are 11 items: resting pulse, GI upset, sweating, tremor, restlessness, yawning, pupil size, anxiety, aches, gooseflesh skin, and runny nose/tearing. Each measure has a different maximum point value depending on observed symptoms.
  Of the participants at baseline, 146 participants in Standard Procedure and 201 participants in Rapid Procedure had COWS assessed in this first admission day. Population: Not all participants who enrolled and participated in baseline data collection had COWS collected on first day of admission (baseline assessments were conducted most frequently after the first day of admission)
  units on a scale
    number analyzed (Participants) | 146 | 201 | 347
    (all) | 5.7 (4.50) | 4.8 (3.53) | 5.2 (3.99)
History of lifetime opioid overdose [Count of Participants; unit: Participants] — Collected via participant self-report
  Participants | 89 | 111 | 200
Number of lifetime overdoses [Mean (Standard Deviation); unit: overdoses] — collected by participant self-report Population: 89 participants in Standard Procedure indicated history of overdose in their lifetime, and 88 of them provided data on the total number of overdoses via self-report (1 missing). 111 participants in Rapid Procedure indicated history of overdose in their lifetime, and all of them provided data on the total number of overdoses via self-reporting (none missing).
  overdoses
    number analyzed (Participants) | 88 | 111 | 199
    (all) | 4.5 (6.92) | 4.1 (4.59) | 4.3 (5.73)
Baseline substance use (Urine Drug Screen) [Number; unit: Number of positive test results] — Urine drug screen results recorded after testing for adulteration and confirming sample is fit for testing. Buprenorphine taper is part of study treatment initiation, and use of benzodiazepines for treatment of withdrawal symptoms was encouraged. Number of positive tests will not match number of participants assessed because UDS categories are not mutually exclusive and participants may have a positive result for one, multiple or no substances.
  Number of positive test results
    Opiates | 38 | 64 | 102
    Oxycodone | 11 | 7 | 18
    Methadone | 7 | 4 | 11
    Buprenorphine | 127 | 129 | 256
    Amphetamine | 36 | 67 | 103
    Barbiturate | 1 | 1 | 2
    Benzodiazepines | 63 | 116 | 179
    Marijuana | 83 | 78 | 161
    Cocaine | 55 | 49 | 104
    Ecstasy (MDMA) | 8 | 7 | 15
    Methamphetamine | 38 | 61 | 99
    Phencyclidine | 3 | 0 | 3
    Fentanyl | 123 | 140 | 263
TLFB substance use (at least once in the past 7 days) [Number; unit: # participants with reported use] — Collected via participant self-report within the defined categories. Participants assessed will not match with reports of drug use as participants may report use of one, multiple, or none of the listed drugs.
  # participants with reported use
    Heavy alcohol use (Females: 3 or more; Males: 4 or more (drinks per day)) | 27 | 28 | 55
    Heroin/Fentanyl | 132 | 151 | 283
    Opioid analgesics | 35 | 37 | 72
    Buprenorphine | 17 | 11 | 28
    Methadone | 6 | 1 | 7
    No opioids (heroin/fentanyl, opioid analgesics, buprenorphine, methadone) | 7 | 12 | 19
    Other amphetamine | 5 | 6 | 11
    Benzodiazepines | 18 | 43 | 61
    Cannabis | 80 | 87 | 167
    Cocaine | 51 | 42 | 93
    Ecstasy (MDMA) | 10 | 4 | 14
    Methamphetamine | 50 | 56 | 106
    Inhalants | 1 | 2 | 3
    Other drugs | 1 | 5 | 6
    Missing | 21 | 29 | 50
TLFB substance use (at least once in the past 30 days) [Number; unit: # participants with reported use] — Collected via participant self-report within the defined categories. Participants assessed will not match with reports of drug use as participants may report use of one, multiple, or none of the listed drugs.
  # participants with reported use
    Heavy alcohol use (Females: 3 or more; Males: 4 or more (drinks per day)) | 36 | 39 | 75
    Heroin/Fentanyl | 141 | 155 | 296
    Opioid analgesics | 45 | 47 | 92
    Buprenorphine | 25 | 16 | 41
    Methadone | 11 | 3 | 14
    No opioids (heroine/fentanyl, opioid analgesics, buprenorphine, methadone) | 2 | 8 | 10
    Other amphetamine | 9 | 10 | 19
    Benzodiazepines | 28 | 64 | 92
    Cannabis | 95 | 114 | 209
    Cocaine | 70 | 61 | 131
    Ecstasy (MDMA) | 18 | 6 | 24
    Methamphetamine | 60 | 73 | 133
    Inhalants | 1 | 2 | 3
    Other drugs | 1 | 6 | 7
    Missing | 21 | 29 | 50
Type of baseline heroin/fentanyl last use from TLFB [Number; unit: # participants with reported use] — Collected via participant self-report within the defined categories. Participants assessed will not match with reports of drug use as participants may report use of one, multiple, or none of the listed drugs.
  # participants with reported use
    No use | 28 | 35 | 63
    Oral | 3 | 1 | 4
    Nasal | 54 | 66 | 120
    Smoking | 25 | 12 | 37
    Injection | 56 | 73 | 129
    Missing | 21 | 29 | 50
Type of baseline prescription opioid last use [Number; unit: # participants with reported use] — Collected via participant self-report within the defined categories. Participants assessed will not match with reports of drug use as participants may report use of one, multiple, or none of the listed drugs.
  # participants with reported use
    Nasal | 18 | 11 | 29
    Smoking | 1 | 1 | 2
    Injection | 5 | 1 | 6
Type of baseline methadone last use [Number; unit: # participants with reported use] — Collected via participant self-report within the defined categories. Participants assessed will not match with reports of drug use as participants may report use of one, multiple, or none of the listed drugs.
  # participants with reported use
    Nasal | 1 | 0 | 1
    Injection | 1 | 0 | 1
Type of baseline buprenorphine last use [Number; unit: # participants with reported use] — Collected via participant self-report within the defined categories. Participants assessed will not match with reports of drug use as participants may report use of one, multiple, or none of the listed drugs.
  # participants with reported use
    Nasal | 0 | 0 | 0
    Injection | 0 | 0 | 0
Substance use disorder [Number; unit: participants] — Categories from DSM-5 study assessment, completed by a physician while assessing participant.
  participants
    Opioid use disorder | 189 | 224 | 413
    Alcohol use disorder | 105 | 111 | 216
    Amphetamine use disorder | 85 | 119 | 204
    Cannabis use disorder | 129 | 159 | 288
    Cocaine use disorder | 109 | 104 | 213
    Sedative use disorder | 68 | 95 | 163

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Who Receive the First XR-NTX Injection (Dichotomous: Did or Did Not Receive First Dose of XR-NTX)
Description: The primary goal of the study is to show RP is non-inferior to SP XR-NTX induction method.
Time Frame: Induction Phase: 1-30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Induction Method | Rapid Induction Method
Number analyzed (Participants) | 190 | 225
Participants | 68 | 141

2. Secondary Outcome: Mean for Time From Admission to First XR-NTX Injection by Treatment Group.
Description: Time to receipt of first injection of XR-NTX from day of admission for participants that receive first injection of XR-NTX.
Time Frame: Induction Phase: 1-30 days
Population: Only participants who received first injection of XR-NTX were analyzed for days to first injection.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard Induction Method | Rapid Induction Method
Number analyzed (Participants) | 68 | 141
Days | 14.5 (3.57) | 7.0 (1.42)

3. Secondary Outcome: Mean of Individual Participant's Opioid Craving Measured by Visual Analog Scales (VAS) During Induction Phase
Description: Craving for opioids measured by Visual Analog Scales (VAS). Scale 0-100, 0 no craving and 100 Most intense craving possible
Time Frame: Induction Phase: 1-30 days
Reporting Status: Not Posted

4. Secondary Outcome: Mean of Individual Participant's Opioid Craving Measured by Visual Analog Scales (VAS) During Post-induction Weeks 1 Through 8
Description: as for outcome 3
Time Frame: Post Induction Phase: 1-8 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Mean of Individual Participant's Opioid Withdrawal Measured by Subjective Opioid Withdrawal Scale (SOWS) During Induction Phase
Description: Opioid withdrawal symptoms as measured by the Subjective Opioid Withdrawal Scale (SOWS). Scale 0-64, with the higher score representing greater withdrawal severity.
Time Frame: Induction Phase: 1-30 days
Reporting Status: Not Posted

6. Secondary Outcome: Mean of Individual Participant's Opioid Withdrawal Measured by Subjective Opioid Withdrawal Scale (SOWS) During Post-induction Weeks 1 Through 4
Description: as for outcome 5
Time Frame: Post Induction Phase: 1 - 4 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Mean of Individual Participant's Opioid Withdrawal Measured by Clinical Opioid Withdrawal Scale (COWS) During Induction Phase
Description: Opioid withdrawal symptoms as measured by the Clinical Opiate Withdrawal Scale (COWS). Scale 0-59, with the higher score representing greater withdrawal severity.
Time Frame: Induction Phase: 1-30 days
Reporting Status: Not Posted

8. Secondary Outcome: Mean of Individual Participant's Opioid Craving Measured by Clinical Opioid Withdrawal Scale (COWS) During Post-induction Weeks 1 Through 4
Description: as for outcome 7
Time Frame: Post Induction Phase: 1 - 4 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Mean for Individual Participant's Patient Health Questionnaire (PHQ-9) Score During Induction Phase
Description: Other depressive, anxiety, and subacute withdrawal symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9). Scale 0-27, with the higher score representing greater severity.
Time Frame: Induction Phase: 1-30 days
Reporting Status: Not Posted

10. Secondary Outcome: Mean for Individual Participant's Patient Health Questionnaire (PHQ-9) Score During Post-induction Weeks 1 Through 8
Description: as for outcome 9
Time Frame: Post Induction Phase: 1 - 8 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Mean for Individual Participant's General Anxiety Disorder (GAD-7) Score During Induction Phase
Description: Other depressive, anxiety, and subacute withdrawal symptoms as measured by the General Anxiety Disorder-7 (GAD-7). Scale 0-21, with the higher score representing greater severity.
Time Frame: Induction Phase: 1-30 days
Reporting Status: Not Posted

12. Secondary Outcome: Mean for Individual Participant's General Anxiety Disorder (GAD-7) Score During Post-induction Weeks 1 Through 8
Description: as for outcome 11
Time Frame: Post Induction Phase: 1 - 8 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Frequency of Targeted Safety Events Related to Study Medication and Any Serious Adverse Events During Induction Period and During Eight Weeks of Post-induction Treatment
Description: Safety, as measured by targeted safety events and serious adverse events.
Time Frame: Induction Phase- 1 - 30 days, Post Induction Phase- 1-8 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Number of Medical Visits and Therapy Completed During Follow up Treatment.
Description: Engagement with medical visits and therapy (based on medical management log, XR- NTX dose log, Psychosocial log).
Time Frame: Post Induction Phase: 1 - 8 weeks
Reporting Status: Not Posted

15. Secondary Outcome: Percent of Patients Reporting Continued Treatment With Medication for Opioid Use Disorder (MOUD) at Week 8
Description: Use of medication for opioid use disorder (MOUD) as measured by patient self-report on Timeline Followback (TLFB).
Time Frame: Post Induction Phase: Week 8
Reporting Status: Not Posted

16. Secondary Outcome: Percent of Participants Positive for Opioids Using Weekly TLFB During Eight Weeks of Post-induction
Description: Opioid abstinence, as measured by the Timeline Followback (TLFB) (self-report days using opioids)
Time Frame: Post Induction Phase: 1 - 8 weeks
Reporting Status: Not Posted

17. Secondary Outcome: Percent of Participants Positive for Opioids Using Urine Drug Screens at Week 4 and 8
Description: Opioid abstinence, as measured by the proportion of opioid-positive urine tests.
Time Frame: Post Induction Phase: Week 4 and Week 8
Reporting Status: Not Posted

18. Secondary Outcome: Percent of Participants Positive for Cocaine, Sedatives, Alcohol, Cannabis, and Tobacco Using Weekly TLFB During Eight Weeks of Post- Induction
Description: Use of alcohol and other drugs of abuse (e.g., cocaine, other stimulants, cannabis, benzodiazepines), by self-report
Time Frame: Post Induction Phase: 1 - 8 weeks
Reporting Status: Not Posted

19. Secondary Outcome: Percent of Participants Positive for Cocaine, Sedatives, Alcohol, Cannabis, and Tobacco Using Urine Drug Screens at Week 4 and 8
Description: Use of alcohol and other drugs of abuse (e.g., cocaine, other stimulants, cannabis, benzodiazepines), by urine drug screens.
Time Frame: Post Induction Phase: Week 4 and Week 8
Reporting Status: Not Posted

20. Secondary Outcome: Proportion of Participants That Receive Second and Third Injection of XR-NTX (at 1 Month and 2 Months, From First Injection)
Description: Retention in the trial to receive the second and the third XR-NTX injections.
Time Frame: Post Induction Phase: Week 4 and Week 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 70 weeks
Arm/Group | Standard Induction Method | Rapid Induction Method
All-Cause Mortality (participants affected / at risk) | 1/190 | 0/225
Serious Adverse Events (participants affected / at risk) | 7/190 | 12/225
Other Adverse Events (participants affected / at risk) | 7/190 | 27/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Induction Method (N=190) | Rapid Induction Method (N=225)
Overdose (Injury, poisoning and procedural complications) | 1 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 2
Suicide Attempt (Psychiatric disorders) | 0 | 1
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Abscess (neck) (Infections and infestations) | 0 | 1
Drug withdrawal convulsions (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Death (General disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Induction Method (N=190) | Rapid Induction Method (N=225)
Fall Event (Injury, poisoning and procedural complications) | 1 | 8
Acute change in mental status (Psychiatric disorders) | 1 | 1
Acute mental complication likely exacerbated by the stress of withdrawal (Psychiatric disorders) | 5 | 13
Acute psychiatric symptoms (Psychiatric disorders) | 0 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT04762537/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT04762537/SAP_001.pdf